CLINICAL TRIAL: NCT01198561
Title: Repetitive Transcranial Magnetic Stimulation(rTMS) in the Treatment of Depression : Effect of TMS on Depression, Cognitive Function, and Regional Cerebral Glucose Metabolism
Brief Title: Repetitive Transcranial Magnetic Stimulation(rTMS) in the Treatment of Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Doh Kwan Kim, M.D., Ph.D. / Professor, Samsung Medical Center
Other Study IDs: 2005-08-072
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Major Depressive Disorder
Keywords: repetitive Transcranial Magnetic Stimulation; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma and DNAs
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- repetitive Transcranial Magnetic Stimulation: repetitive Transcranial Magnetic Stimulation is a depressive patient group treated with rTMS
  Interventions: Device: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — 10 times repetitive TMS, high frequency

SUMMARY:
The objective of this study is to investigate the antidepressant efficacy of rTMS, and to assess cortical metabolism before and after rTMS sessions in patients with major depression. We also aimed to investigate differences between the responders and nonresponders to rTMS and what would predict clinical response to rTMS.

DETAILED DESCRIPTION:
The specific aims of this study is to: (1) evaluate the antidepressant efficacy of rTMS on major depression; (2) evaluate the effects of rTMS on cognitive function in depressive patients; (3) assess the effects of rTMS on cerebral glucose metabolism in depressive patients as measured by 18FDG PET; (4) investigate the differences of the regional cerebral glucose uptake changes during rTMS between responders and nonresponders to rTMS.

ELIGIBILITY:
Inclusion Criteria:

* Twenty patients fulfilling the diagnostic criteria of major depression according to DSM IV will be enrolled in the study.
* Antidepressant medication will be maintained throughout the study period.

Exclusion Criteria:

* Exclusion criteria are current neurological or other psychiatric disorders, as well as a history of epileptic seizures, substantial brain damage or neurosurgical operation, according to established safety criteria.
* To exclude the effect of drug changes on post-rTMS cerebral glucose metabolism, the combinations and dosage of pre-rTMS antidepressant drugs will remain unchanged until the post-rTMS 18FDG PET is done.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with major depressive disorder, who were not responsive to antidepressants
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2006-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Hamilton depression rating scale (HAM-D 17) | baseline, 1, 2, and 4 weeks after TMS
  measuring instrument of severity of depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Doh K KIm, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Kangnam-Ku, South Korea